CLINICAL TRIAL: NCT01691794
Title: A Prospective Single Arm, Open-label, International, Multicenter Study to Evaluate the Safety of Atazanavir (ATV) Capsule Boosted With Ritonavir (RTV) With an Optimized NRTI Background Therapy, in HIV Infected, Antiretroviral Naive and Experienced Pediatric Subjects Greater Than or Equal to 6 Years to Less Than 18 Years
Brief Title: Safety Sudy of Atazanavir Boosted With Ritonavir in the Treatment of HIV Infection in Pediatric Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI424-452; 2011-003300-21 (EudraCT Number)
Record Dates: First submitted 2012-09-21; First posted 2012-09-25 (Estimated); Results first posted 2015-11-30 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2018-03

CONDITIONS: HIV, Pediatric
MeSH Terms: interventions — Atazanavir Sulfate; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Atazanavir, 150 mg + Ritonavir, 100 mg (weight:15 to <20 kg) (Active Comparator): Participants with baseline weight of 15 to <20 kg received 150 mg of atazanavir plus 100 mg of ritonavir once daily with an optimized background therapy of 2 nucleoside reverse transcriptase inhibitors (NRTIs) for 24 weeks. In countries without locally approved pediatric indication for atazanavir, patients may continue to receive study treatment, with regular 12-week visits, until the age of 18 years.
  Interventions: Drug: Atazanavir; Drug: Ritonavir
- Atazanavir, 200 mg + Ritonavir, 100 mg (weight: 20 to <40 kg) (Active Comparator): Participants with baseline weight of 20 to <40 kg received 200 mg of atazanavir plus 100 mg of ritonavir once daily with an optimized background therapy of 2 NRTIs for 24 weeks. In countries without locally approved pediatric indication for atazanavir, patients may continue to receive study treatment, with regular 12-week visits, until the age of 18 years.
  Interventions: Drug: Atazanavir; Drug: Ritonavir
- Atazanavir, 300 mg + Ritonavir, 100 mg (weight: ≥ 40 kg) (Active Comparator): Participants with baseline weight ≥ 40 kg received 300 mg of atazanavir plus 100 mg of ritonavir once daily with an optimized background therapy of 2 NRTIs for 24 weeks. In countries without locally approved pediatric indication for atazanavir, patients may continue to receive study treatment, with regular 12-week visits, until the age of 18 years.
  Interventions: Drug: Atazanavir; Drug: Ritonavir

INTERVENTIONS:
Drug: Atazanavir
  Other Names: Reyataz; BMS-232632
Drug: Ritonavir
  Other Names: Norvir

SUMMARY:
The purpose of this study is to collect safety clinical data in HIV-infected pediatric patients aged 6 and older to younger than18 years and weighing 15 kg or more, who are receiving atazanavir capsule boosted with ritonavir and an optimized nucleoside reverse transcriptase inhibitor backbone therapy as part of their antiretroviral regimen.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HIV-1 infection diagnosed by protocol criteria
* Male or female children, ≥ 6 years to <17 years 6 months of age at the time of first treatment
* Antiretroviral-naïve or treatment-experienced participants with a detectable viral load
* Antiretroviral-naïve participants must have genotypic sensitivity at screening to atazanavir and at least 2 nucleoside reverse transcriptase inhibitors (NRTIs), which have been approved for pediatric use and dosed per local country label
* Antiretroviral-experienced participants must have documented genotypic and phenotypic sensitivity at screening to atazanavir (fold change in susceptibility <2.2) and at least 2 NRTIs, which have been approved for pediatric use and dosed per local country label.

Exclusion Criteria:

* Experienced participants who received atazanavir with or without ritonavir at any time prior to study enrollment
* Antiretroviral-naive or -experienced HIV-1 infected patients with contraindication to study medications
* Documented cardiac conduction abnormality, significant cardiac dysfunction, or a history syncope
* Family history of QTc interval syndrome, Brugada syndrome, right ventricular dysplasia, or a corrected QTc interval of >440 ms at screening
* One of the following cardiac rhythm abnormalities documented on the screening electrocardiogram:

  1. First degree atrioventricular (AV) block, as defined by protocol
  2. Type I second degree AV block while awake, type II second degree AV block at any time, complete AV block at any time, or age-adjusted heart rate <2nd percentile
* Coinfection with either hepatitis B or C virus

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2012-11-30 (Actual); Primary Completion 2014-10-31 (Actual); Study Completion 2017-02-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (21):
- United States (3):
  - Phoenix Children'S Hospital, Phoenix, Arizona
  - Grady Health System Ponce Family And Youth Clinic, Atlanta, Georgia
  - Children'S Medical Center Of Dallas, Dallas, Texas
- Argentina (2):
  - Local Institution, Buenos Aires, Bs As, Buenos Aires
  - Local Institution, Buenos Aires
- Brazil (4):
  - Local Institution, Salvador, Estado de Bahia
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, São Paulo, São Paulo
  - Local Institution, São Paulo
- Local Institution, Santiago, Santiago Metropolitan, Chile
- Mexico (4):
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, Mérida, Yucatán
  - Local Institution, Puebla City
- Local Institution, Lima, Peru
- Russia (2):
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
- South Africa (4):
  - Local Institution, Port Elizabeth, Eastern Cape
  - Local Institution, Bloemfontein, Free State
  - Local Institution, Soweto, Gauteng
  - Local Institution, Cape Town, Western Cape

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Overall, 108 participants were enrolled, and 59 received treatment.
Groups:
- Atazanavir, 150 mg + Ritonavir, 100 mg (Weight: 15 to <20 kg): Participants with baseline weight of 15 to <20 kg received 150 mg of atazanavir in capsule formation plus 100 mg of ritonavir once daily with an optimized background therapy of 2 nucleoside reverse transcriptase inhibitors (NRTIs) for 24 weeks. In countries without locally approved pediatric indication for atazanavir, patients were eligible to receive study treatment, with regular 12-week visits, until the age of 18 years.
- Atazanavir, 200 mg + Ritonavir, 100 mg (Weight: 20 to <40 kg): Participants with baseline weight of 20 to <40 kg received 200 mg of atazanavir plus 100 mg of ritonavir once daily with an optimized background therapy of 2 NRTIs for 24 weeks. In countries without locally approved pediatric indication for atazanavir, patients were eligible to receive study treatment, with regular 12-week visits, until the age of 18 years.
- Atazanavir, 300 mg + Ritonavir, 100 mg (Weight: ≥40 kg): Participants with baseline weight ≥40 kg received 300 mg of atazanavir plus 100 mg of ritonavir once daily with an optimized background therapy of 2 NRTIs for 24 weeks. In countries without locally approved pediatric indication for atazanavir, patients were eligible to receive study treatment, with regular 12-week visits, until the age of 18 years.
Period: Overall Study
Arm/Group | Atazanavir, 150 mg + Ritonavir, 100 mg (Weight: 15 to <20 kg) | Atazanavir, 200 mg + Ritonavir, 100 mg (Weight: 20 to <40 kg) | Atazanavir, 300 mg + Ritonavir, 100 mg (Weight: ≥40 kg)
Started | 3 | 33 | 23
Completed | 2 (Completed baseline to End of Study) | 15 (Completed baseline to End of Study) | 13 (Completed baseline to End of Study)
Not Completed | 1 | 18 | 10
Not completed — Poor/Non-Compliance | 1 | 4 | 1
Not completed — Death | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 7 | 1
Not completed — Participant request to discontinue | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Completed Only first 24 weeks of study | 0 | 2 | 3
Not completed — Did not complete first 24 weeks of study | 0 | 3 | 3

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Atazanavir, 150 mg + Ritonavir, 100 mg (Weight: 15 to <20 kg) | Atazanavir, 200 mg + Ritonavir, 100 mg (Weight: 20 to <40 kg) | Atazanavir, 300 mg + Ritonavir, 100 mg (Weight: ≥40 kg) | Total
Number analyzed (Participants) | 3 | 33 | 23 | 59
Age, Continuous [Mean (Standard Deviation); unit: Years] | 6.0 (0.0) | 10.7 (2.67) | 14.7 (1.72) | 12.0 (3.26)
Age, Customized [Median (Full Range); unit: Years] | 6.0 [6 to 6] | 11.0 [6 to 16] | 15.0 [11 to 17] | 12.0 [6 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 17 | 11 | 30
  Male | 1 | 16 | 12 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 2 | 3
  Not Hispanic or Latino | 1 | 2 | 2 | 5
  Unknown or Not Reported | 2 | 30 | 19 | 51
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 1 | 5 | 4 | 10
  Black/African American | 2 | 24 | 9 | 35
  Other | 0 | 4 | 10 | 14
Region of Enrollment [Number; unit: Participants]
  Africa | 2 | 24 | 8 | 34
  Europe | 0 | 1 | 0 | 1
  North America | 1 | 0 | 3 | 4
  South America | 0 | 8 | 12 | 20
Country [Number; unit: Participants]
  Argentina | 0 | 3 | 0 | 3
  Brazil | 0 | 3 | 4 | 7
  Chile | 0 | 1 | 2 | 3
  Mexico | 1 | 0 | 1 | 2
  Peru | 0 | 1 | 6 | 7
  Russia | 0 | 1 | 0 | 1
  South Africa | 2 | 24 | 8 | 34
  United States | 0 | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Died and With Serious Adverse Events (SAEs), Adverse Events (AEs) Leading to Discontinuation, Grade 2-4 Related AEs, Grade 3-4 AEs, and Centers for Disease Control (CDC) Class C AIDS Events
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Related=having certain, probable, possible, or unknown relationship to study drug. Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, Grade 4=Life-threatening or disabling, Grade 5=Death.
Time Frame: From first dose to last dose plus 30 days (assessed up to February 2017, approximately 42 months)
Population: All participants who received at least 1 dose of study drug
Measure: Number; unit: Participants
Arm/Group | Atazanavir, 150 mg + Ritonavir, 100 mg (Weight: 15 to <20 kg) | Atazanavir, 200 mg + Ritonavir, 100 mg (Weight: 20 to <40 kg) | Atazanavir, 300 mg + Ritonavir, 100 mg (Weight: ≥40 kg)
Number analyzed (Participants) | 3 | 33 | 23
Participants
  Deaths | 0 | 0 | 1
  SAEs | 1 | 3 | 4
  AEs leading to discontinuation | 0 | 1 | 2
  Grade 2-4 related AEs | 1 | 3 | 5
  Grade 3-4 AEs | 0 | 3 | 5
  CDC Class C AIDS events | 0 | 1 | 0

2. Primary Outcome: Number of Participants With Laboratory Test Results Meeting the Criteria for Abnormal, Grades 1-4
Description: Hematocrit (%): Grade (Gr) 1= ≥28.5- <31.5; Gr 2= ≥24- <28.5; Gr 3= ≥19.5- <24; Gr 4= <19.5. Hemoglobin (g/dL): Grade (Gr)1=8.5-10.0; Gr 2=7.5-8.4; Gr 3=6.50-7.4; Gr 4= <6.5. Platelets (/mm^3): Gr 1=100,000-124,999; Gr 2=50,000-99,999; Gr 3=25,000-49,999; Gr 4= <25,000. White blood cells (/mm^3): Gr 1=2000-2500; Gr 2=1500-1999; Gr 3=1000-1499; Gr 4= <1000. Neutrophils (/mm^3): Gr 1=1000-1500; Gr 2= ≥750-1000; Gr 3= ≥500-750; Gr 4= <500. Alanine transaminase (ALT), alkaline phosphatase (ALP), aspartate transaminase (AST) (*upper limit of normal [ULN]): Gr 1=1.5-2.5; Gr 2=2.6-5.0; Gr 3=5.1-10.0; Gr 4= >10.0. Total bilirubin (adult and pediatric >14 days) (*ULN): Gr 1=1.1-1.5; Gr 2=1.6-2.5; Gr 3=2.6-5.0; Gr 4= >5.0. Albumin (g/dL): Gr 1= 3.1- <LLN; Gr 2=2.0-2.9; Gr 3= <2.0; Gr 4=NA. Amylase (*ULN): Gr 1=1.10-1.39; Gr 2=1.40-2.09; Gr 3=2.10-5.0; Gr 4= >5. Lipase (*ULN): Gr 1=1.1-1.5; Gr 2=1.6-3.0; Gr 3=3.1-5.0; Gr 4= >5.0.
Time Frame: After first dose to last dose plus 30 days (assessed up to February 2017, approximately 42 months)
Population: All participants who received at least 1 dose of study drug
Measure: Number; unit: Participants
Arm/Group | Atazanavir, 150 mg + Ritonavir, 100 mg (Weight: 15 to <20 kg) | Atazanavir, 200 mg + Ritonavir, 100 mg (Weight: 20 to <40 kg) | Atazanavir, 300 mg + Ritonavir, 100 mg (Weight: ≥40 kg)
Number analyzed (Participants) | 3 | 33 | 23
Participants
  Hematocrit | 0 | 3 | 0
  Hemoglobin | 0 | 5 | 0
  Platelets | 0 | 0 | 1
  White blood cells | 0 | 3 | 0
  Neutrophils+bands (absolute) | 1 | 13 | 4
  ALT | 1 | 6 | 9
  AST | 0 | 6 | 5
  ALP | 1 | 11 | 12
  Total bilirubin | 3 | 26 | 17
  Albumin | 2 | 15 | 6
  Amylase | 2 | 27 | 14
  Lipase | 0 | 15 | 8

3. Primary Outcome: Number of Participants With Laboratory Test Results Meeting the Criteria for Abnormal, Grades 1-4 (Continued)
Description: Blood urea nitrogen (*upper limit of normal [ULN]): Grade (Gr) 1=1.25-2.5; Gr 2=2.6-5.0; Gr 3=5.1-10; Gr 4= >10. Uric acid (mg/dL): Gr 1=7.5-10.0; Gr 2=10.1-12; Gr 3=12.1-15.0; Gr 4= >15.0. Bicarbonate (mEqL): Gr 1= 19.0-21.0; Gr 2=15.0-18.0; Gr 3=41-45; Gr 4= >45. Calcium, low (mg/dL): Gr 1=7.8-8.4; Gr 2=7.0-7.7; Gr 3=6.1-6.9; Gr 4= <6.1.Potassium (mEq/L), high: Gr 1=5.6-6.0; Gr 2=6.1-6.5; Gr 3=6.6-7.0; Gr 4= >7.0. Potassium (mEq/L), low: Gr 1=3.1-3.4; Gr 2=2.5-2.9; Gr 3=2.0-2.4; Gr 4= <2.0. Sodium (mEq/L), low: Gr 1=130-135; Gr 2=125-129; Gr 3=121-124; Gr 4= <1. Total cholesterol, fasting (mg/dL): Gr 1=200-239; Gr 2=240-300; Gr 3= >300; Gr 4=Not applicable (NA). Low-density lipoprotein (LDL) cholesterol, fasting (mg/dL): Gr 1=130-159; Gr 2=160-190; Gr 3= >190; Gr 4= NA. Glucose, low (mg/dL): Gr 1= 55-64; Gr 2=40-54; Gr 3=30-39; Gr 4= <30. Glucose, fasting (mg/dL): Gr 1=110-125; Gr 2=126-250; Gr 3=251-500; Gr 4 >500.
Time Frame: After first dose to last dose plus 30 days (assessed up to February 2017, approximately 42 months)
Population: All participants who received at least 1 dose of study drug
Measure: Number; unit: Participants
Arm/Group | Atazanavir, 150 mg + Ritonavir, 100 mg (Weight: 15 to <20 kg) | Atazanavir, 200 mg + Ritonavir, 100 mg (Weight: 20 to <40 kg) | Atazanavir, 300 mg + Ritonavir, 100 mg (Weight: ≥40 kg)
Number analyzed (Participants) | 3 | 33 | 23
Participants
  Blood urea nitrogen | 0 | 3 | 0
  Uric acid | 0 | 2 | 3
  Bicarbonate, low | 3 | 29 | 17
  Calcium, low | 0 | 2 | 3
  Potassium, high | 0 | 2 | 1
  Potassium, low | 0 | 2 | 0
  Total cholesterol, fasting (n=3, 31, 21) | 0 | 10 | 6
  Sodium, low | 1 | 13 | 0
  LDL cholesterol, fasting (n=3, 31, 21) | 0 | 7 | 3
  Glucose, low (n=1, 11, 9) | 0 | 3 | 0
  Glucose, fasting, high (3, 31, 22) | 0 | 3 | 1
  Calcium, high | 0 | 2 | 0
  Chloride, high | 0 | 0 | 2
  Chloride, low | 0 | 0 | 0
  Glucose, Non-Fasting, High | 0 | 0 | 0
  Sodium, high | 0 | 1 | 1
  Creatinine | 0 | 1 | 0
  Triglycerides, fasting | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose to last dose plus 30 days (assessed up to February 2017, approximately 42 months)
Groups:
- B/L Weight 15 to Less Than 20 kg: Participants with baseline weight of 15 to <20 kg received 150 mg of atazanavir in capsule formation plus 100 mg of ritonavir once daily with an optimized background therapy of 2 nucleoside reverse transcriptase inhibitors (NRTIs) for 24 weeks. In countries without locally approved pediatric indication for atazanavir, patients were eligible to receive study treatment, with regular 12-week visits, until the age of 18 years.
- B/L Weight 20 to Less Than 40 kg: Participants with baseline weight of 20 to <40 kg received 200 mg of atazanavir plus 100 mg of ritonavir once daily with an optimized background therapy of 2 NRTIs for 24 weeks. In countries without locally approved pediatric indication for atazanavir, patients were eligible to receive study treatment, with regular 12-week visits, until the age of 18 years.
- B/L Weight Greater Than and Equal 40 kg: Participants with baseline weight ≥40 kg received 300 mg of atazanavir plus 100 mg of ritonavir once daily with an optimized background therapy of 2 NRTIs for 24 weeks. In countries without locally approved pediatric indication for atazanavir, patients were eligible to receive study treatment, with regular 12-week visits, until the age of 18 years.
Arm/Group | B/L Weight 15 to Less Than 20 kg | B/L Weight 20 to Less Than 40 kg | B/L Weight Greater Than and Equal 40 kg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/33 | 1/23
Serious Adverse Events (participants affected / at risk) | 1/3 | 3/33 | 4/23
Other Adverse Events (participants affected / at risk) | 3/3 | 26/33 | 20/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | B/L Weight 15 to Less Than 20 kg (N=3) | B/L Weight 20 to Less Than 40 kg (N=33) | B/L Weight Greater Than and Equal 40 kg (N=23)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1
Meningitis bacterial (Infections and infestations) | 0 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0
Abnormal behaviour (Psychiatric disorders) | 0 | 0 | 1
Glomerulonephritis (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Post streptococcal glomerulonephritis (Renal and urinary disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | B/L Weight 15 to Less Than 20 kg (N=3) | B/L Weight 20 to Less Than 40 kg (N=33) | B/L Weight Greater Than and Equal 40 kg (N=23)
Atrioventricular block first degree (Cardiac disorders) | 0 | 3 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 5
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 1
Nausea (Gastrointestinal disorders) | 0 | 2 | 4
Toothache (Gastrointestinal disorders) | 0 | 3 | 0
Vomiting (Gastrointestinal disorders) | 0 | 7 | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 2 | 4
Jaundice (Hepatobiliary disorders) | 1 | 2 | 6
Ocular icterus (Hepatobiliary disorders) | 0 | 1 | 3
Bronchitis (Infections and infestations) | 1 | 2 | 0
Conjunctivitis (Infections and infestations) | 0 | 2 | 2
Gastroenteritis (Infections and infestations) | 1 | 3 | 0
Impetigo (Infections and infestations) | 0 | 1 | 2
Influenza (Infections and infestations) | 1 | 3 | 3
Nasopharyngitis (Infections and infestations) | 1 | 3 | 6
Oral herpes (Infections and infestations) | 0 | 4 | 1
Otitis media (Infections and infestations) | 1 | 2 | 2
Tonsillitis (Infections and infestations) | 1 | 4 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 13 | 4
Headache (Nervous system disorders) | 0 | 4 | 2
Depression (Psychiatric disorders) | 0 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 9 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 4 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 4 | 2
Ear pain (Ear and labyrinth disorders) | 0 | 2 | 0
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 2 | 0
Pyrexia (General disorders) | 0 | 2 | 0
Abscess (Infections and infestations) | 0 | 2 | 0
Pharyngitis (Infections and infestations) | 1 | 1 | 0
Pharyngotonsillitis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.